CLINICAL TRIAL: NCT03718546
Title: Identifying Predictors of Poor Health-Related Quality-of-Life Among Pediatric Hematopoietic Stem Cell Donors
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 17-SIBS
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (6):
- Sibling pediatric donors: Donors who are donating to a sibling
- Sibling recipients and caregivers: Recipients who are receiving a transplant from a sibling
- Non-donor sibling: From the donor-recipient families
- Non-donor siblings: Of patients receiving unrelated transplants
- Healthy comparison: A matched sample
- Parents: Parent/caregiver of study participating donor.

SUMMARY:
To compare donors to their non-donor counterparts and healthy controls as well as to generate trajectory classes based on longitudinal patterns of donor HRQoL and identify predictors of poor donor HRQoL.

DETAILED DESCRIPTION:
There is limited data to show the effects that donation has on pediatric donors to their siblings. There is widespread agreement that it is critical to investigate the medical and psychosocial aspects of sibling pediatric HSC donation for multiple reasons including (a) the vulnerability of the pediatric population undergoing donation, (b) increasing use of pediatric HSC donation as a therapeutic option, (c) evidence that ~20% of pediatric HSC donors experience clinically important HRQoL deficits, and (d) the impact that improved understanding of factors predicting poor HRQoL will have on our ability to develop guidelines and/or interventions for assisting at-risk donors/families. The proposed study will help to compare donors to their non-donor counterparts and healthy controls as well as to generate trajectory classes based on longitudinal patterns of donor HRQoL and identify predictors of poor donor HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* Participants must fall into one of the following categories:

  * Donor between the age of 5 and 17 who is donating to a sibling
  * Parent/caregiver of study participating donor
  * Recipient sibling aged 5 to 17 of study participating donor
  * Any of the donor's non-donor/non-recipient siblings between 5 and 17
  * Any child between 5 and 17 with a brother or sister (also between 5 and 17) receiving a transplant from an unrelated source
* Be willing and able to provide signed informed consent:

  * Adults must give consent for their children's and, if applicable, their own participation
  * Assent will be obtained in accordance with guidelines at the participant's transplant institution
* Be willing and able to respond to psychological assessment questions
* Must be the donor's first donation
* Recipient must consent to the CIBMTR research database

Exclusion Criteria:

* For families with pediatric donors aged 5 to 17, at minimum, the donor child and/or one parent must consent/assent to participation. If that minimum is not met, the family will be excluded
* Donor or non-donor siblings who do not live in the same household as the recipient at lease half of the time
* Unable to consent/assent or complete a phone interview in English

  * Parents may consent/assent in Spanish
* No access to a telephone

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric donors, their recipients and caregivers, non-donor siblings from the donor-recipient families, and non-donor siblings of patients receiving unrelated transplants.
Sampling Method: Non-Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-10-08 (Actual)

PRIMARY OUTCOMES:
HRQoL (Health Related Quality of Life) | 1 year
  To longitudinally and quantitatively describe the HRQoL of a diverse nation-wide cohort of sibling pediatric Hematopoietic Stem Cell (HSC) donors (Peripheral Blood Stem Cell or Bone Marrow) and to compare their HRQoL to that of (1) healthy non-donor sibling from the same family, (2) siblings of children with similar diseases who receive alternate treatments (e.g., unrelated cord blood transplants), and (3) healthy age, gender, and race/ethnicity-matched controls.

SECONDARY OUTCOMES:
1 year post-donation | 1 year
  To identify and examine donor HRQoL trajectories from pre- through 1 year post-donation.
Donor characteristics | 1 year
  To determine which donor characteristics (e.g., demographic, psychosocial, and donation-related), recipient characteristics (e.g., recipient disease, transplant complications and outcomes), family characteristics (e.g., composition, cohesiveness, stress), and transplant center characteristics (e.g., presence of a donor advocate) most strongly predict membership in trajectory classes with poor HRQoL among donors.

CONTACTS AND LOCATIONS:
Overall Officials: Galen Switzer, Ph.D, Principal Investigator — University of Pittsburgh
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - Loma Linda University, Loma Linda, California
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale New Haven Hospital, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Niklaus Children's Hospital, Miami, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Louisville Hospital - James Brown Cancer Center, Louisville, Kentucky
  - Children's Hospital of New Orleans/LSUHSC, New Orleans, Louisiana
  - NIH/NCI, Bethesda, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - The Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Westchester Medical Center, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Children's Health (formerly Children's Medical Center Dallas), Dallas, Texas
  - Methodist Healthcare System of San Antonio/Texas Transplant Institute, San Antonio, Texas
  - University of Utah Blood and Marrow Transplant Program - Pediatrics, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No